CLINICAL TRIAL: NCT03418051
Title: Neuromuscular Mechanisms of Manual Therapies in Chronic Ankle Instability Patients
Brief Title: Mechanisms of Manual Therapies in CAI Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 17-2655; 1R21AT009704-01 (NIH)
Record Dates: First submitted 2018-01-24; First posted 2018-02-01 (Actual); Results first posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-07

CONDITIONS: Ankle Inversion Sprain; Chronic Instability of Joint
Keywords: Ankle Instability; Manual Therapy; Massage; Ankle Joint Mobilization; Biomechanics; Neuromuscular
MeSH Terms: interventions — Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Control group that will receive no intervention throughout the duration of the study (2-weeks).
- Joint Mobilization (Experimental): Participants will receive 6, 5-minute treatment sessions over 2-weeks. Each session will consist of 2, 2-minute bouts of Grade III anterior-to-posterior talocrural joint mobilization with 1-minute between sets. Mobilizations will be large-amplitude, 1-s rhythmic oscillations from the mid- to end range of arthrokinematic motion.
  Interventions: Other: Joint Mobilization
- Massage (Experimental): Participants will receive 6, 5-minute treatment sessions over 2-weeks. Each session will consist of 2, 2-minute bouts of plantar massage bouts with 1-minute between sets. The massage will be a combination of petrissage and effleurage to the entire plantar surface.
  Interventions: Other: Massage

INTERVENTIONS:
Other: Joint Mobilization — Participants will receive 6, 5-minute treatment sessions over 2-weeks. Each session will consist of 2, 2-minute bouts of Grade II anterior to posterior ankle joint mobilizations with 1-minute between sets. Mobilizations will be large-amplitude, 1-s rhythmic oscillations from the mid- to end range of arthrokinematic motion.
  Other Names: Ankle Joint Mobilization
  Arms: Joint Mobilization
Other: Massage — Participants will receive 6, 5-minute treatment sessions over 2-weeks. Each session will consist of 2, 2-minute bouts of plantar massage with 1-minute between sets. The massage will be a combination of petrissage and effleurage to the entire plantar surface.
  Other Names: Plantar Massage
  Arms: Massage

SUMMARY:
ABSTRACT:

Injury associated with sport and recreation is a leading reason for physical activity cessation, which is linked with significant long-term negative consequences. Lateral ankle sprains are the most common injuries associated with physical activity and at least 40% of individuals who sprain their ankle will go on to develop chronic ankle instability (CAI), a multifaceted condition linked with life-long residual symptoms and post-traumatic ankle osteoarthritis. Our long term goal is to develop intervention strategies to decrease disability associated with acute and chronic ankle injury and prevent posttraumatic ankle osteoarthritis. Conventional rehabilitation strategies, are only moderately successful because they ignore the full spectrum of residual symptoms associated with CAI. Manual therapies such as ankle joint mobilizations and plantar massage target sensory pathways not addressed by conventional treatments and have been shown to improve patient-reported outcomes, dorsiflexion range of motion, and postural control in CAI patients. While these early results are promising, the underlying neuromuscular mechanisms of these manual therapies remain unknown. Therefore the objective of this R21 proposal is to determine the neuromuscular mechanisms underlying the improvements observed following independent ankle joint mobilization and plantar massage interventions in CAI patients. To comprehensively evaluate the neuromuscular mechanisms of the experimental treatments, baseline assessments of peripheral (ankle joint proprioception, light-touch detection thresholds, spinal (H-Reflex of the soleus and fibularis longus), and supraspinal mechanisms (cortical activation, cortical excitability, and cortical mapping, sensory organization) will be assessed. Participants will then be randomly assigned to receive ankle joint mobilizations (n=20), plantar massage (n=20), or a control intervention (n=20) which will consist of 6, 5-minute treatments over 2-weeks. Post-intervention assessments will be completed within 48-hours of the final treatment session. Separate ANOVAs will assess the effects of treatment group (ankle joint mobilization, plantar massage, control) and time (baseline, post-treatment) on peripheral, spinal, and supraspinal neuromuscular mechanisms in CAI participants. Associations among neuromuscular mechanisms and secondary measures (biomechanics and postural control) will also be assessed. The results of this investigation will elucidate multifaceted mechanisms of novel and effective manual therapies (ankle joint mobilizations and plantar massage) in those with CAI.

ELIGIBILITY:
Inclusion criteria:

Individuals with Chronic Ankle Instability which will be defined as those individuals who:

* have sustained at least two lateral ankle sprains;
* have experienced at least one episode of giving way within the past 6-months;
* answer 4 or more questions of "yes" on the Ankle Instability Instrument;
* have self-assessed disability scores of ≤90% on the Foot and Ankle Ability Measure;
* have self-assessed disability scores ≤80% on the Foot and Ankle Ability Measure-Sport.

Exclusion criteria for Chronic Ankle Instability will include:

* known vestibular and vision problems,
* acute lower extremities and head injuries (<6 weeks),
* chronic musculoskeletal conditions known to affect balance (e.g., Anterior Cruciate Ligament deficiency) and
* a history of ankle surgeries to fix internal derangement.

Participants will also be excluded if they have any of the following which are contraindications to Transcranial Magnetic Stimulation testing:

* metal anywhere in the head (except in the mouth),
* pacemakers,
* implantable medical pumps,
* ventriculo-peritoneal shunts,
* intracardiac lines,
* history of seizures,
* history of stroke
* history of serious head trauma.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Wikstrom, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Fetzer Hall, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The entire dataset will link the outcomes and demographics but will be devoid of patient identifying information. Upon completion of the study, this information will be available to those who request the data, meet the access criteria, and agree to a data use agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available following completion of the study for two years.
Access Criteria: Data will be made available to other investigators that contact the PI and provide written commitment (i.e. data use agreement) to: 1) only use the data for purposes currently unplanned by the principal investigators or co-investigators; 2) only use the data for research purposes and not to contact patients or potential future research subjects; 3) securing the data using appropriate computer technology; as well as 4) destroying or returning the data following completion of data analysis.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Joint Mobilization | Massage
Started | 20 | 20 | 20
Completed | 14 | 18 | 17
Not Completed | 6 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Joint Mobilization | Massage | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.5 (.8) | 21.9 (3.9) | 20.9 (3.2) | 20.7 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 12 | 20
  Male | 15 | 17 | 8 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 2 | 7
  Not Hispanic or Latino | 18 | 17 | 18 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 5
  White | 15 | 17 | 14 | 46
  More than one race | 1 | 0 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 20 | 60
Ankle Instability Instrument [Mean (Standard Deviation); unit: units on a scale] — The ankle instability instrument (AII) is a questionnaire used to capture self-reported data from the participant regarding history of ankle injury and perceived deficits in function. The outcome is the number of 'yes' responses to the questions asked.
  Minimum = 0 Maximum = 9 Higher scores = greater perceived disability.
  units on a scale | 7.4 (1.35) | 7.4 (1.46) | 7.0 (1.23) | 7.3 (1.34)
Number of ankle sprains [Mean (Standard Deviation); unit: sprains] | 4.5 (3.5) | 4.25 (2.35) | 5.1 (3.85) | 4.6 (3.27)
Number of giving way episodes [Mean (Standard Deviation); unit: giving way episodes] — A giving way episode is defined as an episode where the participant had the sensation that their ankle was about to give way but such an event did not result in a recurrent ankle sprain. The outcome is the number of giving way episodes within the past 6 months.
  giving way episodes | 7 (1.56) | 10.4 (16.13) | 9.15 (8.63) | 8.85 (11.2)
Outcome Expectations for Exercise Scale [Mean (Standard Deviation); unit: units on a scale] — The Outcome Expectations for Exercise Scale was used to determine if participants believe that receiving a manual therapy treatment would result in a positive outcome. This was captured via a single question using a Likert scale (range: 1 to 5). Higher scores indicate a higher perception that a manual therapy treatment would result in a positive outcome.
  units on a scale | 2.8 (0.83) | 2.8 (0.76) | 2.9 (0.85) | 2.83 (0.81)

OUTCOME MEASURES:

1. Primary Outcome: ML COP Velocity From Baseline to Post Intervention
Description: % Modulation of ML COP velocity.
  First, center of pressure (COP) is calculated in the mediolateral (ML) direction [side to side] with eyes open and closed. COP velocity represents the average speed at which an individual's COP moves during the 10 second single limb stance trial.
  Next, % modulation is calculated. This estimates the weight given to visual information during eyes open stance based on the magnitude of change in ML COP Velocity that occurs when vision is removed relative to the eyes open condition (control condition). The following formula is used: % Modulation = (eyes closed balance score - eyes open balance score) / eyes open balance score. Positive scores indicate a greater reliance on visual information as ML COP velocity increased when eyes were closed relative to the eyes open condition. A ML COP velocity change greater than the eyes open value would result in a value >100%. This analysis focused on baseline to the immediate post-treatment assessment.
Time Frame: Baseline and 24-72 hours post intervention
Population: All missing data was the result of participants being lost to follow-up.
Measure: Mean (Standard Deviation); unit: % modulation
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 18 | 19 | 19
% modulation
  Baseline | 119.91 (47.38) | 118.91 (47.38) | 121.07 (44.55)
  Post Intervention | 116.99 (36.16) | 128.23 (40.10) | 121.20 (42.83)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.824, ANOVA — A priori alpha level was set to 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.426, ANOVA — A priori alpha level was set to 0.05

2. Primary Outcome: ML COP Velocity From Baseline to Follow-Up
Description: % Modulation of ML COP velocity.
  First, center of pressure (COP) is calculated in the mediolateral (ML) direction [side to side] with eyes open and closed. COP velocity represents the average speed at which an individual's COP moves during the 10 second single limb stance trial.
  Next, % modulation is calculated. This estimates the weight given to visual information during eyes open stance based on the magnitude of change in ML COP Velocity that occurs when vision is removed relative to the eyes open condition (control condition). The following formula is used: % Modulation = (eyes closed balance score - eyes open balance score) / eyes open balance score. Positive scores indicate a greater reliance on visual information as ML COP velocity increased when eyes were closed relative to the eyes open condition. A ML COP velocity change greater than the eyes open value would result in a value >100%. This analysis focused on baseline to the Follow-Up assessment.
Time Frame: Baseline and 4-week Follow-Up
Population: All missing data was the result of participants being lost to follow-up.
Measure: Mean (Standard Deviation); unit: % modulation
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 14 | 18 | 17
% modulation
  Baseline | 119.71 (48.70) | 116.13 (41.37) | 119.14 (46.66)
  Follow-Up | 118.86 (45.11) | 110.80 (46.45) | 111.06 (43.86)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.722, ANOVA — A priori alpha level was set to 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.843, ANOVA — A priori alpha level was set to 0.05

3. Primary Outcome: AP COP Velocity From Baseline to Post Intervention
Description: % Modulation of AP COP velocity.
  First, center of pressure (COP) is calculated in the anterioposterior (AP) direction [front to back]. COP velocity represents the average speed at which an individual's COP moves during the 10 second single limb stance trial.
  Next, % modulation is calculated. This estimates the weight given to visual information during eyes open stance based on the magnitude of change in ML COP Velocity that occurs when vision is removed relative to the eyes open condition (control condition). The following formula is used: % Modulation = (eyes closed balance score - eyes open balance score) / eyes open balance score. Positive scores indicate a greater reliance on visual information as ML COP velocity increased when eyes were closed relative to the eyes open condition. A ML COP velocity change greater than the eyes open value would result in a value >100%. This analysis focused on baseline to the immediate post-treatment assessment.
Time Frame: Baseline and 24-72 hours post intervention
Population: All missing data was the result of participants being lost to follow-up.
Measure: Mean (Standard Deviation); unit: % modulation
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 18 | 19 | 19
% modulation
  Baseline | 117.40 (31.73) | 115.84 (47.32) | 126.50 (37.95)
  Post Intervention | 120.91 (33.69) | 122.51 (39.05) | 100.91 (38.53)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.046, ANOVA — A priori alpha level was set to 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.845, ANOVA — A priori alpha level was set to 0.05

4. Primary Outcome: AP COP Velocity From Baseline to Follow-up
Description: % Modulation of AP COP velocity.
  First, center of pressure (COP) is calculated in the anterioposterior (AP) direction [front to back] with eyes open and closed. COP velocity represents the average speed at which an individual's COP moves during the 10 second single limb stance trial.
  Next, % modulation is calculated. This estimates the weight given to visual information during eyes open stance based on the magnitude of change in ML COP Velocity that occurs when vision is removed relative to the eyes open condition (control condition). The following formula is used: % Modulation = (eyes closed balance score - eyes open balance score) / eyes open balance score. Positive scores indicate a greater reliance on visual information as ML COP velocity increased when eyes were closed relative to the eyes open condition. A ML COP velocity change greater than the eyes open value would result in a value >100%. This analysis focused on baseline to the follow-up assessment.
Time Frame: Baseline and 4-week Follow-Up
Population: All missing data was the result of participants being lost to follow-up.
Measure: Mean (Standard Deviation); unit: % modulation
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 14 | 18 | 17
% modulation
  Baseline | 119.48 (33.02) | 116.69 (48.19) | 123.93 (39.40)
  Follow-Up | 117.67 (40.04) | 105.10 (48.54) | 97.96 (35.18)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.138, ANOVA — A priori alpha level was set to 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.523, ANOVA — A priori alpha level was set to 0.05

5. Primary Outcome: ML TTB From Baseline to Post Intervention
Description: % Modulation of ML Time-to-Boundary.
  First, time-to-Boundary (TTB) is calculated in the mediolateral (ML) direction [side to side] with eyes open and closed. TTB represents the time (s) it would take for a participant's center of pressure (i.e. vertical projection of the center of mass) to reach their base of support (i.e. boundary) based on the instantaneous position and velocity of the center of pressure. The base of support is represents the length and width of an individual's foot.
  Next, % modulation is calculated. This estimates the weight given to visual information during eyes open stance based on the magnitude of change in ML TTB that occurs when vision is removed relative to the eyes open condition (control condition). The following formula is used: % Modulation = (eyes open balance score - eyes closed balance score) / eyes open balance score. Negative scores indicate a greater reliance on visual information as ML TTB decreased with eyes closed.
Time Frame: Baseline and 24-72 hours post intervention
Population: All missing data was the result of participants being lost to follow-up.
Measure: Mean (Standard Deviation); unit: % modulation
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 18 | 19 | 19
% modulation
  Baseline | -50.76 (13.41) | -54.97 (8.98) | -55.41 (10.81)
  Post Intervention | -55.99 (7.14) | -56.61 (10.43) | -52.28 (11.73)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.069, ANOVA — A priori alpha level was set to 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.413, ANOVA — A priori alpha level was set to 0.05

6. Primary Outcome: ML TTB From Baseline to Follow-Up
Description: as for outcome 5
Time Frame: Baseline and 4-week Follow-Up
Population: Missing data was due to participants lost to follow up.
Measure: Mean (Standard Deviation); unit: % modulation
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 14 | 18 | 17
% modulation
  Baseline | -48.98 (14.31) | -54.18 (9.41) | -51.12 (13.00)
  Follow-Up | -51.12 (13.00) | -52.18 (12.69) | -53.12 (10.91)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.604, ANOVA — A priori alpha level was set to 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.499, ANOVA — A priori alpha level was set to 0.05

7. Primary Outcome: AP TTB From Baseline to Post Intervention
Description: % Modulation of AP Time-to-Boundary.
  First, time-to-Boundary (TTB) is calculated in the anterioposterior (AP) direction [front to back] with eyes open and closed. TTB represents the time (s) it would take for a participant's center of pressure (i.e. vertical projection of the center of mass) to reach their base of support (i.e. boundary) based on the instantaneous position and velocity of the center of pressure. The base of support is represents the length and width of an individual's foot.
  Next, % modulation is calculated. This estimates the weight given to visual information during eyes open stance based on the magnitude of change in AP TTB that occurs when vision is removed relative to the eyes open condition (control condition). The following formula is used: % Modulation = (eyes open balance score - eyes closed balance score) / eyes open balance score. Negative scores indicate a greater reliance on visual information as AP TTB decreased with eyes closed.
Time Frame: Baseline and 24-72 hours post intervention
Population: All missing data was the result of participants being lost to follow-up.
Measure: Mean (Standard Deviation); unit: % modulation
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 18 | 18 | 19
% modulation
  Baseline | -52.54 (9.67) | -54.59 (8.81) | -57.53 (8.24)
  Post Intervention | -52.97 (7.31) | -54.39 (11.01) | -48.81 (8.67)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.005, ANOVA — A priori threshold was set at 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.853, ANOVA — A priori threshold set at 0.05

8. Primary Outcome: AP TTB From Baseline to Follow-Up
Description: % Modulation of AP Time-to-Boundary.
  First, time-to-Boundary is calculated in the anterioposterior (AP) direction [front to back] with eyes open and closed. Time-to-boundary represents the time (s) it would take for a participant's center of pressure (i.e. vertical projection of the center of mass) to reach their base of support (i.e. boundary) based on the instantaneous position and velocity of the center of pressure. The base of support is represents the length and width of an individual's foot.
  Next, % modulation is calculated. This estimates the weight given to visual information during eyes open stance based on the magnitude of change in AP TTB that occurs when vision is removed relative to the eyes open condition (control condition). The following formula is used: % Modulation = (eyes open balance score - eyes closed balance score) / eyes open balance score. Negative scores indicate a greater reliance on visual information as AP TTB decreased with eyes closed.
Time Frame: Baseline and 4-week Follow-Up
Population: All missing data was the result of participants being lost to follow-up.
Measure: Mean (Standard Deviation); unit: % modulation
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 14 | 18 | 17
% modulation
  Baseline | -52.95 (10.40) | -55.09 (8.36) | -53.98 (10.53)
  Follow-Up | -51.94 (11.40) | -47.38 (12.05) | -48.81 (9.92)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.142, ANOVA — A priori threshold set to 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.167, ANOVA — A priori threshold set at 0.05

9. Primary Outcome: 95% Confidence Ellipse From Baseline to Post Intervention
Description: % Modulation of 95% Confidence Ellipse.
  First, center of pressure (COP) excursion [movement] is calculated and the magnitude of an ellipse that contains 95% of all data points is calculated with eyes open and closed. The resulting outcome is calculated from a 10 second single limb stance trial.
  Next, % modulation is calculated. This estimates the weight given to visual information during eyes open stance based on the magnitude of change that occurs when vision is removed relative to the eyes open condition (control condition). The following formula is used: % Modulation = (eyes closed balance score - eyes open balance score) / eyes open balance score. Positive scores indicate a greater reliance on visual information as the variable increased when eyes were closed relative to the eyes open condition. A change greater than the eyes open value would result in a value >100%. This analysis focused on baseline to the immediate post-treatment assessment.
Time Frame: Baseline and 24-72 hours post intervention
Population: All missing data was the result of participants being lost to follow-up.
Measure: Mean (Standard Deviation); unit: % modulation
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 18 | 18 | 19
% modulation
  Baseline | 270.91 (168.28) | 270.91 (168.28) | 290.70 (128.07)
  Post-Intervention | 267.85 (127.60) | 283.26 (111.89) | 275.92 (142.78)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.849, ANOVA — A priori alpha set at 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.993, ANOVA — A priori threshold set at 0.05

10. Primary Outcome: 95% Confidence Ellipse From Baseline to Follow-Up
Description: as for outcome 9
Time Frame: Baseline and 4-week Follow-Up
Population: All missing data was the result of participants being lost to follow-up.
Measure: Mean (Standard Deviation); unit: % modulation
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 14 | 18 | 17
% modulation
  Baseline | 286.29 (173.43) | 272.07 (142.18) | 282.06 (129.60)
  Follow-Up | 317.46 (146.05) | 254.06 (165.90) | 267.92 (134.57)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.535, ANOVA — A priori alpha level was set to 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.569, ANOVA — A priori alpha level was set to 0.05

11. Secondary Outcome: Plantar Flexion Joint Position Sense From Baseline to Post Intervention
Description: Amount of error, measured in degrees, from a target angle of plantar flexion. Participants are shown a target ankle and asked to replicate that angle (i.e. joint position) with their eyes closed. The amount of error from the target angle is recorded as the joint position sense. Larger values (i.e. greater error) indicates worse joint position sense. This analysis focused on baseline to the immediate post-treatment assessment.
Time Frame: Baseline and 24-72 hours post intervention
Population: All missing data was the result of participants being lost to follow-up.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 19 | 20 | 19
Degrees
  Baseline | 3.00 (1.82) | 3.25 (1.60) | 3.73 (2.54)
  Post Intervention | 2.22 (1.36) | 1.97 (1.54) | 2.42 (1.67)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.405, ANOVA — A priori threshold was 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.229, ANOVA — A priori threshold set to 0.05

12. Secondary Outcome: Plantar Flexion Joint Position Sense From Baseline to Follow-Up
Description: Amount of error, measured in degrees, from a target angle of plantar flexion. Participants are shown a target ankle and asked to replicate that angle (i.e. joint position) with their eyes closed. The amount of error from the target angle is recorded as the joint position sense. Larger values (i.e. greater error) indicates worse joint position sense. This analysis focused on baseline to the follow-up assessment.
Time Frame: Baseline and 4-week Follow-Up
Population: Missing data was due to participants being lost to follow up.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 14 | 18 | 18
Degrees
  Baseline | 3.04 (1.78) | 3.04 (1.78) | 3.72 (2.61)
  Follow-Up | 2.35 (1.95) | 1.51 (1.49) | 2.62 (2.20)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.609, ANOVA — A priori threshold set at 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.027, ANOVA — A priori threshold was set at 0.05

13. Secondary Outcome: 1st Metatarsal Light-touch Threshold From Baseline to Post Intervention
Description: Minimal amount of pressure that can be detected by an individual at the head of the 1st metatarsal. Semmes-Weinstein monofilaments, of different diameters (mm), are pressed against the skin using an established 4-2-1 stepping algorithm. Higher values (thresholds) indicate worse light touch sensation thresholds. his analysis focused on baseline to the immediate post-treatment assessment.
Time Frame: Baseline and 24-72 hours post intervention
Population: Missing data due to participants being lost at follow up.
Measure: Median (Standard Deviation); unit: mm
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 18 | 20 | 19
mm
  Baseline | 2.83 (0.62) | 3.22 (0.55) | 3.61 (0.76)
  Post intervention | 3.41 (0.57) | 3.22 (0.73) | 2.83 (0.54)
Statistical Analysis 1: Comparison: Control vs Joint Mobilization vs Massage; Test type: Superiority; p = 0.613, Independent sample Mann-Whitney U — A priori alpha set at 0.05

14. Secondary Outcome: 1st Metatarsal Light-touch Threshold From Baseline to Follow-Up
Description: Minimal amount of pressure that can be detected by an individual at the head of the 1st metatarsal. Semmes-Weinstein monofilaments, of different diameters (mm), are pressed against the skin using an established 4-2-1 stepping algorithm. Higher values (thresholds) indicate worse light touch sensation thresholds. This analysis focused on baseline to the follow-up assessment.
Time Frame: Baseline and 4-week Follow-Up
Population: Missing data due to participants being lost at follow up.
Measure: Median (Standard Deviation); unit: mm
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 14 | 18 | 18
mm
  Baseline | 2.95 (0.67) | 3.22 (0.57) | 3.41 (0.77)
  Follow-Up | 3.22 (0.67) | 3.22 (0.58) | 2.83 (0.81)
Statistical Analysis 1: Comparison: Control vs Joint Mobilization vs Massage; Test type: Superiority; p = 0.925, Independent sample Mann-Whitney U — A priori threshold set at 0.05

15. Secondary Outcome: 5th Metatarsal Light-touch Threshold From Baseline to Post Intervention
Description: Minimal amount of pressure that can be detected by an individual at the base of the 5th metatarsal. Semmes-Weinstein monofilaments, of different diameters (mm), are pressed against the skin using an established 4-2-1 stepping algorithm. Higher values (thresholds) indicate worse light touch sensation thresholds. This analysis focused on baseline to the immediate post-treatment assessment.
Time Frame: Baseline and 24-72 hours post intervention
Population: Missing data due to participants being lost at follow up.
Measure: Median (Standard Deviation); unit: mm
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 18 | 20 | 19
mm
  Baseline | 3.22 (0.60) | 3.22 (0.59) | 3.84 (0.75)
  Post Intervention | 3.61 (0.69) | 3.41 (0.23) | 3.22 (0.69)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.641, Wilcoxon (Mann-Whitney) — A priori threshold set at 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.897, Wilcoxon (Mann-Whitney) — A priori threshold set at 0.05

16. Secondary Outcome: 5th Metatarsal Light-touch Threshold From Baseline to Follow-Up
Description: Minimal amount of pressure that can be detected by an individual at the base of the 5th metatarsal. Semmes-Weinstein monofilaments, of different diameters (mm), are pressed against the skin using an established 4-2-1 stepping algorithm. Higher values (thresholds) indicate worse light touch sensation thresholds. This analysis focused on baseline to the follow-up assessment.
Time Frame: Baseline and 4-week Follow Up
Population: Missing data due to participants being lost at follow up.
Measure: Median (Standard Deviation); unit: mm
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 14 | 18 | 18
mm
  Baseline | 3.22 (0.62) | 3.22 (0.61) | 3.84 (0.76)
  Follow-Up | 3.61 (0.50) | 3.41 (0.85) | 3.61 (0.91)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.561, Wilcoxon (Mann-Whitney) — A priori threshold set at 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.925, Wilcoxon (Mann-Whitney) — A priori threshold set at 0.05

17. Secondary Outcome: Soleus H:M Ratio From Baseline to Post Intervention
Description: This measure shows the percentage of excited alpha motor neurons (H) within a muscle upon electrical stimulation, relative to the total number of alpha motor neurons in the same muscle (M). Higher scores represent a greater percentage of excitability (i.e. activation) and is thought to represent better function of the spinal motor pathway. This analysis focused on baseline to the immediate post-treatment assessment.
  The test is performed using an electric stimulator and electromyography (EMG) to record muscle responses. Stimulation intensity is increased on sequential trials to capture both the H-wave and M-wave responses.
Time Frame: Baseline and 24-72 hours post intervention
Population: Missing data due to participants being lost to follow up or technical issues with equipment.
Measure: Mean (Standard Deviation); unit: H:M Ratio
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 18 | 19 | 15
H:M Ratio
  Baseline | 0.68 (.140) | 0.65 (0.18) | 0.63 (0.30)
  Post-Intervention | 0.67 (0.14) | 0.62 (0.12) | 0.64 (0.29)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.233, ANOVA — A priori threshold set at 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.634, ANOVA — A priori threshold set at 0.05

18. Secondary Outcome: Soleus H:M Ratio From Baseline to Follow-Up
Description: as for outcome 17
Time Frame: Baseline and 4-week Follow-Up
Population: Missing data due to participants being lost to follow up or technical issues with equipment.
Measure: Mean (Standard Deviation); unit: H:M Ratio
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 14 | 17 | 13
H:M Ratio
  Baseline | 0.67 (0.15) | 0.63 (0.18) | 0.65 (0.25)
  Follow-Up | 0.64 (0.13) | 0.62 (0.16) | 0.67 (0.15)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.233, ANOVA — A priori threshold set at 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.634, ANOVA — A priori threshold set at 0.05

19. Secondary Outcome: Fibularis Longus H:M Ratio From Baseline to Post Intervention
Description: as for outcome 17
Time Frame: Baseline and 24-72 hours post intervention
Population: Missing data due to participants being lost to follow up or technical issues with equipment.
Measure: Mean (Standard Deviation); unit: H:M Ratio
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 18 | 19 | 15
H:M Ratio
  Baseline | 0.34 (0.13) | 0.29 (0.20) | 0.25 (0.20)
  Post-Intervention | 0.27 (0.08) | 0.23 (0.12) | 0.28 (0.17)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.030, ANOVA — A priori threshold set at 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.618, ANOVA — A priori threshold set at 0.05

20. Secondary Outcome: Fibularis Longus H:M Ratio From Baseline to Follow-Up
Description: as for outcome 17
Time Frame: Baseline and 4-week Follow-Up
Population: Missing data due to participants being lost to follow up or technical issues with equipment.
Measure: Mean (Standard Deviation); unit: H:M Ratio
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 14 | 17 | 13
H:M Ratio
  Baseline | 0.30 (0.08) | 0.28 (0.20) | 0.28 (0.20)
  Follow-Up | 0.29 (0.14) | 0.23 (0.11) | 0.32 (0.18)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.456, ANOVA — A priori threshold set at 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.568, ANOVA — A priori threshold set to 0.05

21. Secondary Outcome: Fibularis Longus Active Motor Threshold From Baseline to Post Intervention
Description: A measure of cortical excitability using transcranial electromagnetic stimulation. A higher active motor threshold (AMT) indicates decreased excitability, as a greater stimulus intensity is required to elicit a motor evoke potential (MEP). This analysis focused on baseline to the immediate post-treatment assessment.
Time Frame: Baseline and 24-72 hours post intervention
Population: Missing data due to participants being lost to follow up or technical issues with equipment.
Measure: Mean (Standard Deviation); unit: % maximum intensity
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 16 | 18 | 10
% maximum intensity
  Baseline | 44 (9.87) | 38.38 (8.60) | 40.8 (42.2)
  Post-Intervention | 45.12 (8.37) | 38.27 (6.75) | 42.2 (8.46)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.919, ANOVA — A priori alpha level was set to 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.558, ANOVA — A priori alpha level was set to 0.05

22. Secondary Outcome: Fibularis Longus Active Motor Threshold From Baseline to Follow-Up
Description: as for outcome 21
Time Frame: Baseline and 4-week Follow-Up
Population: Missing data due to participants lost to follow up or technical issues with equipment.
Measure: Mean (Standard Deviation); unit: % maximum intensity
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 12 | 15 | 9
% maximum intensity
  Baseline | 44 (10.23) | 39.6 (8.47) | 41.22 (6.90)
  Follow-Up | 44.75 (9.16) | 40.26 (9.26) | 42.55 (43.80)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.796, ANOVA — A priori alpha level was set to 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.558, ANOVA — A priori alpha level was set to 0.05

23. Secondary Outcome: Cortical Silent Period From Baseline to Post Intervention
Description: A measure of corticospinal inhibition using transcranial electromagnetic stimulation. The cortical silent period (CSP) will be measured as the distance from the end of the motor evoked potential (MEP) to a return of the mean electromyographic (EMG) signal plus two times the standard deviation of the baseline (pre-stimulus) EMG signal. A longer CSP indicates a greater corticospinal inhibition. This analysis focused on baseline to the immediate post-treatment assessment.
Time Frame: Baseline and 24-72 hours post intervention
Population: Missing data due to participants lost to follow up or technical issues with equipment.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 16 | 18 | 10
ms
  Baseline | 0.107 (0.077) | 0.125 (0.084) | 0.122 (0.027)
  Post-Intervention | 0.085 (0.036) | 0.114 (0.038) | 0.091 (0.024)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.701, ANOVA — A priori alpha level was set to 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.68, ANOVA — A priori alpha level was set to 0.05

24. Secondary Outcome: Cortical Silent Period From Baseline to Follow-Up
Description: A measure of corticospinal inhibition using transcranial electromagnetic stimulation. The cortical silent period (CSP) will be measured as the distance from the end of the motor evoked potential (MEP) to a return of the mean electromyographic (EMG) signal plus two times the standard deviation of the baseline (pre-stimulus) EMG signal. A longer CSP indicates a greater corticospinal inhibition. This analysis focused on baseline to the follow-up assessment.
Time Frame: Baseline and 4-week Follow-Up
Population: Missing data due to participants lost to follow up or technical issues with equipment.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 12 | 15 | 9
ms
  Baseline | 0.088 (0.037) | 0.121 (0.087) | 0.114 (0.032)
  Follow Up | 0.088 (0.024) | 0.096 (0.024) | 0.110 (0.046)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.883, ANOVA — A priori threshold set at 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.401, ANOVA — A priori threshold set at 0.05

25. Secondary Outcome: Corticomotor Map Area From Baseline to Post Intervention
Description: A measure representing the size of a muscle's cortical representation using transcranial electromagnetic stimulation. Map area is the number of stimulus positions whose stimulation evoked an average motor evoked potential ≥ the motor evoked potential threshold. An increase would suggest an expansion of the cortical representation of a selected muscle. This analysis focused on baseline to the immediate post-treatment assessment.
Time Frame: Baseline and 24-72 hours post intervention
Population: Missing data due to participants lost to follow up or technical issues with equipment.
Measure: Mean (Standard Deviation); unit: number of positions
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 16 | 18 | 10
number of positions
  Baseline | 13.43 (10.6) | 19.6 (12.0) | 21.8 (15.3)
  Post-Intervention | 16.68 (11.47) | 21.55 (11.4) | 20.2 (12.14)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.393, ANOVA — A priori threshold set at 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.779, ANOVA — A priori threshold set at 0.05

26. Secondary Outcome: Corticomotor Map Area From Baseline to Follow-Up
Description: A measure representing the size of a muscle's cortical representation using transcranial electromagnetic stimulation. Map area is the number of stimulus positions whose stimulation evoked an average motor evoked potential ≥ the motor evoked potential threshold. An increase would suggest an expansion of the cortical representation of a selected muscle. This analysis focused on baseline to the follow-up assessment.
Time Frame: Baseline and 4-week Follow-Up
Population: Missing data due to participants lost at follow-up or technical issues with equipment.
Measure: Mean (Standard Deviation); unit: number of positions
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 12 | 15 | 9
number of positions
  Baseline | 14.3 (11.79) | 16.73 (10.1) | 20.0 (12.92)
  Follow Up | 9.08 (6.17) | 16.73 (6.73) | 20.66 (12.92)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.246, ANOVA — A priori threshold set at 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.191, ANOVA — A priori threshold set at 0.05

27. Secondary Outcome: Corticomotor Map Volume From Baseline to Post Intervention
Description: A measure representing the size of a muscle's cortical representation using transcranial electromagnetic stimulation. Map volume will be calculated as the sum of the mean normalized MEPs recorded with an increase suggesting greater cortical excitability. This analysis focused on baseline to the immediate post-treatment assessment.
Time Frame: Baseline and 24-72 hours post intervention
Population: Missing data due to participants lost to follow up or technical issues with equipment.
Measure: Mean (Standard Deviation); unit: number of positions
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 16 | 18 | 10
number of positions
  Baseline | 0.89 (0.29) | 1.2 (0.60) | 1.07 (0.72)
  Post-Intervention | 0.80 (0.36) | 0.93 (0.23) | 1.05 (0.89)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.703, ANOVA — A priori threshold set at 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.282, ANOVA — A priori threshold set at 0.05

28. Secondary Outcome: Corticomotor Map Volume From Baseline to Follow-Up
Description: measure representing the size of a muscle's cortical representation using transcranial electromagnetic stimulation. Map volume will be calculated as the sum of the mean normalized MEPs recorded with an increase suggesting greater cortical excitability. This analysis focused on baseline to the immediate post-treatment assessment.
Time Frame: Baseline and 4-week Follow-Up
Population: Missing data due to participants lost at follow-up or technical issues with equipment.
Measure: Mean (Standard Deviation); unit: number of positions
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 12 | 15 | 9
number of positions
  Baseline | 0.91 (0.32) | 1.12 (0.62) | 0.99 (0.50)
  Follow-Up | 0.66 (0.39) | 0.74 (0.16) | 0.72 (0.35)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.925, ANOVA — A priori alpha level was set to 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.551, ANOVA — A priori alpha level was set to 0.05

29. Secondary Outcome: Alpha Power Spectral Density From Baseline to Post Intervention
Description: A measure of cortical activation using electroencephalography. Power spectral density (PSD) reflects the distribution of signal power over frequency (micro Volts). Higher PSDs indicate more cortical activity within the alpha bandwidth. This analysis focused on baseline to the immediate post-treatment assessment.
Time Frame: Baseline and 24-72 hours post intervention
Population: Missing data due to participants lost to follow up or technical issues with equipment.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 18 | 20 | 18
mV
  Baseline | 0.739 (0.479) | 0.911 (0.686) | 0.755 (0.428)
  Post Intervention | 0.731 (0.477) | 0.990 (0.887) | 0.633 (0.272)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.506, ANOVA — A priori threshold set at 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.753, ANOVA — A priori threshold at 0.05

30. Secondary Outcome: Alpha Power Spectral Density From Baseline to Follow-Up
Description: A measure of cortical activation using electroencephalography. Power spectral density (PSD) reflects the distribution of signal power over frequency (micro Volts). Higher PSDs indicate more cortical activity within the alpha bandwidth. This analysis focused on baseline to the immediate follow-up assessment.
Time Frame: Baseline and 4-week Follow-Up
Population: Missing data due to participants lost at follow up or technical issues with equipment.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 14 | 16 | 17
mV
  Baseline | 0.669 (0.373) | 0.896 (0.673) | 0.707 (0.425)
  Follow-Up | 0.718 (0.398) | 0.805 (0.471) | 0.701 (0.441)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.777, ANOVA — A priori threshold set at 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.475, ANOVA — A priori threshold set at 0.05

31. Secondary Outcome: Beta Power Spectral Density From Baseline to Post Intervention
Description: A measure of cortical activation using electroencephalography. Power spectral density (PSD) reflects the distribution of signal power over frequency (micro Volts). Higher PSDs indicate more cortical activity within the beta bandwidth. This analysis focused on baseline to the immediate post-treatment assessment.
Time Frame: Baseline and 24-72 hours post intervention
Population: Missing data due to participants lost to follow up or technical issues with equipment.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 18 | 20 | 18
mV
  Baseline | 0.355 (0.147) | 0.480 (0.285) | 0.361 (0.200)
  Post Intervention | 0.336 (0.125) | 0.600 (0.330) | 0.354 (0.162)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.738, ANOVA — A priori threshold set at 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.042, ANOVA — A priori threshold set at 0.05

32. Secondary Outcome: Beta Power Spectral Density From Baseline to Follow-Up
Description: A measure of cortical activation using electroencephalography. Power spectral density (PSD) reflects the distribution of signal power over frequency (micro Volts). Higher PSDs indicate more cortical activity within the beta bandwidth. This analysis focused on baseline to the follow-up assessment.
Time Frame: Baseline and 4-week Follow-Up
Population: Missing data due to participants lost at follow up or technical issues with equipment.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 14 | 16 | 17
mV
  Baseline | 0.310 (0.104) | 0.442 (0.169) | 0.338 (0.206)
  Follow-Up | 0.309 (0.080) | 0.429 (0.169) | 0.311 (0.140)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.738, ANOVA — A priori threshold set at 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.830, ANOVA — A priori threshold set at 0.05

33. Secondary Outcome: Gamma Power Spectral Density From Baseline to Post Intervention
Description: A measure of cortical activation using electroencephalography. Power spectral density (PSD) reflects the distribution of signal power over frequency (micro Volts). Higher PSDs indicate more cortical activity within the gamma bandwidth. This analysis focused on baseline to the immediate post-treatment assessment.
Time Frame: Baseline and 24-72 hours post intervention
Population: Missing data due to participants lost to follow up or technical issues with equipment.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 18 | 20 | 18
mV
  Baseline | 0.116 (0.046) | 0.155 (0.063) | 0.123 (0.052)
  Post Intervention | 0.123 (0.041) | 0.172 (0.097) | 0.125 (0.047)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.700, ANOVA — A priori threshold set at 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.492, ANOVA — A priori threshold set at 0.05

34. Secondary Outcome: Gamma Power Spectral Density From Baseline to Follow-Up
Description: A measure of cortical activation using electroencephalography. Power spectral density (PSD) reflects the distribution of signal power over frequency (micro Volts). Higher PSDs indicate more cortical activity within the gamma bandwidth. This analysis focused on baseline to the follow-up assessment.
Time Frame: Baseline and 4-week Follow-Up
Population: Missing data due to participants lost at follow up or technical issues with equipment.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Control | Joint Mobilization | Massage
Number analyzed (Participants) | 14 | 16 | 17
mV
  Baseline | 0.109 (0.029) | 0.149 (.062) | 0.120 (0.048)
  Follow-Up | 0.116 (0.036) | 0.166 (0.072) | 0.123 (0.041)
Statistical Analysis 1: Comparison: Control vs Massage; Test type: Superiority; p = 0.820, ANOVA — A priori threshold set at 0.05
Statistical Analysis 2: Comparison: Control vs Joint Mobilization; Test type: Superiority; p = 0.526, ANOVA — A priori threshold set at 0.05

35. Other Pre Specified Outcome: Walking Ankle Dorsiflexion at Baseline
Description: Dorsiflexion angle of the ankle at initial contact while walking.
Time Frame: Baseline
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Walking Ankle Dorsiflexion Immediately Post Intervention
Description: Dorsiflexion angle of the ankle at initial contact while walking.
Time Frame: 24-72 hours post intervention
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Walking Ankle Dorsiflexion at 4-weeks Post Intervention
Description: Dorsiflexion angle of the ankle at initial contact while walking.
Time Frame: 4-weeks post intervention
Reporting Status: Not Posted

38. Other Pre Specified Outcome: Walking Loading Rate at Baseline
Description: Rate of weight acceptance while walking
Time Frame: Baseline
Reporting Status: Not Posted

39. Other Pre Specified Outcome: Walking Loading Rate Immediately Post Intervention
Description: Rate of weight acceptance while walking
Time Frame: 24-72 hours post intervention
Reporting Status: Not Posted

40. Other Pre Specified Outcome: Walking Loading Rate at 4-weeks Post Intervention
Description: Rate of weight acceptance while walking
Time Frame: 4-weeks post intervention
Reporting Status: Not Posted

41. Other Pre Specified Outcome: Landing Ankle Dorsiflexion at Baseline
Description: Dorsiflexion angle of the ankle at initial contact while landing from a jump
Time Frame: Baseline
Reporting Status: Not Posted

42. Other Pre Specified Outcome: Landing Ankle Dorsiflexion Immediately Post Intervention
Description: Dorsiflexion angle of the ankle at initial contact while landing from a jump
Time Frame: 24-72 hours post intervention
Reporting Status: Not Posted

43. Other Pre Specified Outcome: Landing Ankle Dorsiflexion at 4-weeks Post Intervention
Description: Dorsiflexion angle of the ankle at initial contact while landing from a jump
Time Frame: 4-weeks post intervention
Reporting Status: Not Posted

44. Other Pre Specified Outcome: Landing Loading Rate at Baseline
Description: Rate of weight acceptance while landing from a jump
Time Frame: Baseline
Reporting Status: Not Posted

45. Other Pre Specified Outcome: Landing Loading Rate Immediately Post Intervention
Description: Rate of weight acceptance while landing from a jump
Time Frame: 24-72 hours post intervention
Reporting Status: Not Posted

46. Other Pre Specified Outcome: Landing Loading Rate at 4-weeks Post Intervention
Description: Rate of weight acceptance while landing from a jump
Time Frame: 4-weeks post intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the Baseline assessment through the Follow-up visit, a total of up to approximately 6 weeks.
Arm/Group | Control | Joint Mobilization | Massage
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT03418051/Prot_SAP_ICF_000.pdf